CLINICAL TRIAL: NCT04429022
Title: Multimodal Pain Management After Robotic-Assisted Total Laparoscopic Hysterectomy
Acronym: RA-TLH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Sarah Andres, D.O., Principal Investigator, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004549
Record Dates: First submitted 2020-04-28; First posted 2020-06-11 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: Hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Acetaminophen; Celecoxib; Ketorolac; Ketorolac Tromethamine; Anesthesia, Obstetrical; Ropivacaine; Anesthetics, Local; Hydromorphone; Oxycodone

STUDY DESIGN:
Intervention Model Description: Prospective cohort with retrospective controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective cohort (Experimental): Pre-Op:
  * Gabapentin 600mg PO PO x 1 prior to surgery (in pre-op)
  * Acetaminophen 1000mg PO x1 prior to surgery (in pre-op)
  Intra-Op:
  * Paracervical block with local anesthetic (0.5% ropivacaine); 10 mL bilaterally (2 point) for total of 20mL
  * Local anesthetic (0.5% ropivacaine) at all laparoscopic port sites; another 10mL
  * Will operate at <15mmHg intra-abdominal pressure, with goal of <12mmHg
  * At end of procedure during closure of fascia, give 30mg ketorolac IV x 1
  Post-Op:
  * Gabapentin 300mg PO BID for 7 days
  * Acetaminophen 1000mg PO q6h x 2 days then 1000mg q6h PRN
  * Celecoxib 200mg PO q 12h x 7d
  * Dilaudid 1mg IV PRN q3h while inpatient; oxycodone 12 x 5mg upon discharge (90MME) if patient did not use any opioids postoperatively while inpatient, will not prescribe opioid medication upon discharge
  Interventions: Drug: Gabapentin; Drug: Acetaminophen; Drug: Celecoxib; Drug: Ketorolac; Procedure: Paracervical block with ropivacaine; Procedure: Local anesthetic injection with ropivacaine at abdominal laparoscopic port sites; Drug: Hydromorphone; Drug: Oxycodone
- Historical Control (Active Comparator): Traditional post-operative opioid medication regimen: Dilaudid 1mg IV PRN q3h while inpatient; Percocets 12 x 5mg/325 (90MME) upon discharge
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Gabapentin — 600mg PO PO x 1 prior to surgery (in pre-op) 300mg PO BID for 7 days post op
  Arms: Prospective cohort
Drug: Acetaminophen — Acetaminophen 1000mg PO x1 prior to surgery (in pre-op) Acetaminophen 1000mg PO q6h x 2 days then 1000mg q6h PRN post op
  Other Names: Tylenol
  Arms: Prospective cohort
Drug: Celecoxib — Celecoxib 200mg PO q 12h x 7d post op
  Other Names: Celebrex
  Arms: Prospective cohort
Drug: Ketorolac — 30mg IV once at end of hysterectomy procedure
  Other Names: Toradol
  Arms: Prospective cohort
Procedure: Paracervical block with ropivacaine — 0.5% ropivacaine; 10 mL bilaterally (2 point) for total of 20mL
  Arms: Prospective cohort
Procedure: Local anesthetic injection with ropivacaine at abdominal laparoscopic port sites — 0.5% ropivacaine; at all laparoscopic port sites; another 10mL ropivacaine in total
  Arms: Prospective cohort
Drug: Hydromorphone — 1mg IV PRN q3h, post op, while inpatient
  Other Names: Dilaudid
Drug: Oxycodone — To be discharged home with: 12 tabs of 5mg PRN q4h
  Arms: Prospective cohort

SUMMARY:
Hysterectomy is the most common major gynecologic surgery performed in the US and is performed for a variety of indications including malignancy, pelvic mass, endometriosis, leiomyoma, and pelvic organ prolapse. The traditional regimen for pain control post-operatively is opioid-based however in light of the opioid epidemic, a transition to non-opioid pain medication regimens is desired by both physicians and patients alike. The goal of this study is to develop a multimodal non-opioid pain medication regimen that minimizes postoperative opioid use after robotic assisted total laparoscopic hysterectomy. Historical controls from January, 2017 to January, 2020 will be compared to our treatment arm from November, 2020 to November, 2022. Included in our treatment protocol is paracervical block and local ropivacaine at abdominal incision sites at surgical start, gabapentin and acetaminophen preoperatively and postoperatively, and celecoxib postoperatively. Opioid use will be measured 0-3 h postop and 3-24h postop (as surrogate marker of time spent recovering in the Post Anesthesia Care Unit (PACU), and during the full length of hospital stay); pain scores will additionally be measured.

DETAILED DESCRIPTION:
Material and Methods:

This is a prospective cohort study with historical controls. Cases of those receiving a non-opioid multimodal pain regimen will be compared to historical controls of those receiving a traditional opioid pain regimen. All patients undergoing robotic total laparoscopic hysterectomy, with or without bilateral salpingo-oophorectomy, with a uterine weight ≤325 grams will be included in this study. Multimodal pain regimen will include the following:

Protocol:

Pre-Op: - Gabapentin 600mg PO PO x 1 prior to surgery (in pre-op area)

* Acetaminophen 1000mg PO x1 prior to surgery (in pre-op area)

Intra-Op:

* Paracervical block with local anesthetic (0.5% ropivacaine); 10 mL bilaterally (2 point) for total of 20mL
* Local anesthetic (0.5% ropivacaine) at all laparoscopic port sites; another 10mL
* Will operate at <15mmHg intra-abdominal pressure with goal of <12mmHg
* At end of procedure during closure of fascia, give 30mg ketorolac IV x 1

Post-Op:

* Gabapentin 300mg PO BID for 7 days
* Acetaminophen 1000mg PO q6h x 2 days then 1000mg q6h PRN
* Celecoxib 200mg PO q 12h x 7d
* Dilaudid 1mg IV PRN q3h while inpatient; oxycodone 12 tabs x 5mg upon discharge (90MME)
* if patient did not use any opioids postoperatively while inpatient, will not prescribe opioid medication upon discharge
* Also include standard post-op medications such as zofran, reglan, mylicon…

Our primary outcome is opioid pain medication needed after surgery. Our secondary outcomes include pain scores as rated subjectively by the patient, length of stay in hours and whether the patient returns to the clinic or emergency department due to post operative pain within a 2 week period.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing robotic-assisted total laparoscopic hysterectomy, with or without bilateral salpingo-oophorectomy
* Uterine weight ≤325 grams

Exclusion Criteria:

* contraindication to any study medications (h/o gastric bypass, gastric ulcers, CKD)
* current opioid prescription

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Andres, D.O., Principal Investigator — University at Buffalo
Locations (1):
- Millard Fillmore Suburban Hospital, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers

REFERENCES:
- [Background] Adajar, A. (2018). 73: Eliminating post-operative narcotic use after mini-laparoscopic hysterectomy: Effectiveness of a multimodal pain management regimen adopted into clinical practice. American Journal of Obstetrics and Gynecology, 218(2), S937-S938. https://doi.org/10.1016/j.ajog.2017.12.092
- [Background] Blanton E, Lamvu G, Patanwala I, Barron KI, Witzeman K, Tu FF, As-Sanie S. Non-opioid pain management in benign minimally invasive hysterectomy: A systematic review. Am J Obstet Gynecol. 2017 Jun;216(6):557-567. doi: 10.1016/j.ajog.2016.12.175. Epub 2016 Dec 30. PMID 28043841
- [Background] Chopra, V., Kown, D., & Sangha, R. (2018). Decreasing Postoperative Narcotic Use for Patients Undergoing Hysterectomy. Journal of Minimally Invasive Gynecology, 25(7), S194-S194. https://doi.org/10.1016/j.jmig.2018.09.526
- [Background] Mark J, Argentieri DM, Gutierrez CA, Morrell K, Eng K, Hutson AD, Mayor P, Szender JB, Starbuck K, Lynam S, Blum B, Akers S, Lele S, Paragh G, Odunsi K, de Leon-Casasola O, Frederick PJ, Zsiros E. Ultrarestrictive Opioid Prescription Protocol for Pain Management After Gynecologic and Abdominal Surgery. JAMA Netw Open. 2018 Dec 7;1(8):e185452. doi: 10.1001/jamanetworkopen.2018.5452. PMID 30646274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the intervention arm, patients were recruited from November 24, 2020 to May 24, 2022. Data for the retrospective controls who underwent their hysterectomy from 11/27/2018 to 12/12/2019, was obtained via chart review. This was a prospective cohort study with retrospective controls. To allow for adjustment to this new protocol, 11 months were allocated to the institution and staff, prior to enrolling patients in the intervention arm.
Pre-assignment Details: 49 patients were analyzed as 18 of 28 intervention arm participants did not receive the intervention or their care required deviation from the from study protocol (e.g., no minimally invasive hysterectomy due to laparotomy, no paracervical block due to indocyanine green injection for lymph node mapping, no postoperative protocol medications due to limited resources and logistical issues). One of the 40 control participants was excluded due to uterine weight exceeding the study protocol range.
Groups:
- Prospective Cohort: Pre-Op:
  * Gabapentin 600mg PO x 1 and
  * Acetaminophen 1000mg PO x1 prior to surgery (in pre-op)
  Intra-Op:
  * Paracervical block with 0.5% ropivacaine; 10 mL bilaterally (2 points), total of 20mL
  * 0.5% ropivacaine subcutaneous injection at all laparoscopic port sites; another 10mL
  * Operate at <15mmHg intra-abdominal pressure, with goal of <12mmHg
  * At end of procedure during closure of fascia, give 30mg ketorolac IV x 1
  Post-Op:
  * Gabapentin 300mg PO BID for 7 days
  * Acetaminophen 1000mg PO q6h x 2 days then 1000mg q6h PRN
  * Celecoxib 200mg PO q 12h x 7d
  * Dilaudid 1mg IV PRN q3h while inpatient; oxycodone 12 x 5mg upon discharge (90MME). If patient did not use any opioids postoperatively while inpatient, will not prescribe opioid medication upon discharge
Period: Overall Study
Arm/Group | Prospective Cohort | Historical Control
Started | 28 | 40
Completed | 10 | 39
Not Completed | 18 | 1
Not completed — Protocol Violation | 18 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Cohort | Historical Control | Total
Number analyzed (Participants) | 10 | 39 | 49
Age, Continuous [Mean (Full Range); unit: years] | 44.60 [32 to 57] | 44.13 [25 to 67] | 44.37 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 39 | 49
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 39 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Pain Medications Required 0-3h Post op in Morphine Milligram Equivalents (MME)
Description: Total opioid pain medications required 0-3h post op in morphine milligram equivalents (MME)
Time Frame: 0-3 hours after surgery
Measure: Mean (Full Range); unit: morphine milligram equivalents (MME)
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
morphine milligram equivalents (MME) | 2.00 [0 to 8.0] | 5.32 [0 to 17.5]

2. Primary Outcome: Total Opioid Pain Medications Required Through 3-24h Post op in MME
Description: Total opioid pain medications required through 3-24h post op in MME
Time Frame: 3-24 hours after surgery
Measure: Mean (Full Range); unit: morphine milligram equivalents (MME)
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
morphine milligram equivalents (MME) | .20 [0 to 2.0] | 12.27 [0 to 52.0]

3. Secondary Outcome: Pain Scores
Description: Subjective, Score 0-10 with 0 being no pain and 10 being severe pain
Time Frame: 3-24 hours after surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
score on a scale | 1.75 [0 to 6.0] | 5.43 [0 to 8.0]

4. Secondary Outcome: Pain Scores
Description: Subjective, Score 0-10 with 0 being no pain and 10 being severe pain
Time Frame: 0-3 hours after surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
score on a scale | 3.82 [0 to 8.0] | 5.13 [0 to 9.0]

5. Secondary Outcome: Length of Stay in Hours
Description: Length of stay in hours
Time Frame: 0- 240 hours
Measure: Mean (Full Range); unit: hours
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
hours | 12.05 [6.0 to 34.0] | 35.82 [10.0 to 239.0]

6. Secondary Outcome: Number of Patients With Return to the Clinic, Emergency Department Due to Post Operative Pain Within a 2 Week Period
Description: Number of patients with return to the clinic, emergency department due to post operative pain within a 2 week period
Time Frame: 0-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
Participants | 1 | 3

7. Secondary Outcome: Operative Time
Description: minutes
Time Frame: 0-300 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
minutes | 128.80 [90 to 179] | 139.69 [73 to 262]

8. Secondary Outcome: Estimated Blood Loss
Description: milliliters (mL)
Time Frame: 0-300 minutes
Measure: Mean (Full Range); unit: milliliters
Arm/Group | Prospective Cohort | Historical Control
Number analyzed (Participants) | 10 | 39
milliliters | 63.50 [10 to 150] | 58.46 [5 to 200]

ADVERSE EVENTS:
Time Frame: 14 days
Description: All participants were assessed for adverse events
Arm/Group | Prospective Cohort | Historical Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/39
Other Adverse Events (participants affected / at risk) | 0/10 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04429022/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT04429022/ICF_002.pdf